CLINICAL TRIAL: NCT00093366
Title: Therapy of Advanced Stage Myelodysplastic Syndrome (MDS) With Arsenic Trioxide Given in Combination With Etanercept: A Phase I/II Study
Brief Title: Arsenic Trioxide and Etanercept in Treating Patients With Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1888.00; FHCRC-1888.00; CDR0000380742 (Registry Identifier: PDQ)
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; myelodysplastic/myeloproliferative disease, unclassifiable; atypical chronic myeloid leukemia; chronic myelomonocytic leukemia
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Myeloproliferative Disorders; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Chronic | interventions — Etanercept; Arsenic Trioxide

INTERVENTIONS:
Biological: etanercept
Drug: arsenic trioxide

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as arsenic trioxide, work in different ways to stop cancer cells from dividing so they stop growing or die. Biological therapies such as etanercept may interfere with the growth of the cancer cells. Combining chemotherapy with biological therapy may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects of giving arsenic trioxide together with etanercept and to see how well it works in treating patients with myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the frequency of hematologic response in patients with intermediate-2 or high-risk myelodysplastic syndromes (MDS) treated with arsenic trioxide and etanercept.
* Determine the efficacy of this regimen in patients with intermediate-1 or low-risk MDS that was refractory to anti-thymocyte globulin and etanercept on protocol FHCRC-1872.
* Correlate results of ex vivo and in vitro studies of phenotypic, cytogenetic, and functional disease characteristics with in vivo treatment response in patients treated with this regimen.
* Determine parameters that are associated with a high probability of disease response in patients treated with this regimen.

OUTLINE: This is a pilot study.

Patients receive arsenic trioxide IV over 1-4 hours on days 1-5 of week 1 and then twice weekly on weeks 2-12 during course 1 (twice weekly on weeks 1-12 during course 2). Patients also receive etanercept subcutaneously twice weekly during weeks 1, 2, 5, 6, 9, and 10. Treatment repeats every 12 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed for 3 months.

PROJECTED ACCRUAL: A total of 15-32 patients will be accrued for this study within 8-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of myelodysplastic syndromes (MDS) meeting 1 of the following criteria:

  * Intermediate-2 or high-risk disease
  * Intermediate-1 or low-risk disease that was refractory to anti-thymocyte globulin and etanercept on protocol FHCRC-1872
* Not eligible for stem cell transplantation for any of the following reasons:

  * Suitable bone marrow donor is not available
  * Ineligible for a transplantation protocol
  * Not willing to undergo transplantation

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 500/mm^3

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* No evidence of cardiac arrhythmia
* No evidence of congestive heart failure
* QTc interval ≤ 460 msec

Pulmonary

* No pneumonia

Other

* Potassium > 4.0 mEq/L (supplemental electrolytes allowed)
* Magnesium > 1.8 mg/dL (supplemental electrolytes allowed)
* No history of anaphylactic reaction to arsenic trioxide
* No active severe infection (e.g., septicemia) within the past 2 weeks
* No other severe disease that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior hematopoietic stem cell transplantation
* More than 4 weeks since prior hematopoietic growth factors for MDS
* More than 4 weeks since prior immunomodulatory therapy for MDS
* No concurrent hematopoietic growth factors for MDS
* No other concurrent immunomodulatory therapy for MDS

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 4 weeks since prior cytotoxic therapy for MDS
* More than 4 weeks since prior experimental therapy for MDS
* No other concurrent cytotoxic therapy for MDS
* No other concurrent experimental therapy for MDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2004-06; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Hematologic response in patients with intermediate-2 or high-risk myelodysplastic syndromes
Efficacy of this regimen in patients with intermediate-1 or low-risk MDS that was refractory to anti-thymocyte globulin and etanercept on protocol FHCRC-1872
Correlate results of ex vivo and in vitro studies on phenotypic, cytogenetic, and functional disease characteristics with in vivo treatment responses
Parameters that are associated with a high probability of response

CONTACTS AND LOCATIONS:
Overall Officials: Bart L. Scott, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States